CLINICAL TRIAL: NCT03472495
Title: Oral vs Intravenous Diltiazem for Rapid Atrial Fibrillation/Flutter Trial
Acronym: OVID RAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20009559
Record Dates: First submitted 2018-02-23; First posted 2018-03-21 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation and Flutter
Keywords: Diltiazem; Atrial Fibrillation; Atrial Flutter; Emergency Medicine
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Immediate Release Diltiazem (Active Comparator): Diltiazem immediate release 60mg orally once (Diltiazem oral product)
  Interventions: Drug: Diltiazem Oral Product
- Continuous Infusion IV Diltiazem (Active Comparator): Diltiazem 2.5-5 mg/hour intravenous Titrate by 1.25 mg every 15-60 minutes. Maximum titration dose 15 mg/hour. Titration Goal of HR <110 (Diltiazem Injectable Product)
  Interventions: Drug: Diltiazem Injectable Product

INTERVENTIONS:
Drug: Diltiazem Oral Product — Diltiazem Immediate Release 60 MG PO Q6H (30 MG PO Q6H if patient is <60 kg)
  Arms: Oral Immediate Release Diltiazem
Drug: Diltiazem Injectable Product — Diltiazem Continuous Infusion Titrated
  Arms: Continuous Infusion IV Diltiazem

SUMMARY:
The primary objective of this study is to compare the incidence of rate control (defined as: HR <110 beats/min or conversion to sinus rhythm) at 2 hours after medication administration between oral immediate release diltiazem and intravenous continuous infusion diltiazem.

DETAILED DESCRIPTION:
Atrial fibrillation (AF), a supraventricular tachyarrhythmia, is the primary diagnosis for over 467,000 hospitalizations each year. Historically, there have been two approaches to managing AF in the emergency department (ED): rate control and rhythm control.

The AFFIRM trial compared rate and rhythm control in 4,060 patients. It found no difference in mortality with the rate control approach and less hospitalizations. As a result, both rhythm and rate control are options in stable patients with an AF duration of < 48 hours. After 48 hours, rate control is preferred because of the increased risk of ischemic stroke. The subsequent RACE II trial, established that lenient heart rate control (HR <110 beats/min) was as effective as strict control (HR <80 beats/min) in preventing cardiovascular events and required less outpatient visits to achieve the goal HR. As a result of both the AFFIRM and RACE II trials, a rate control approach with a goal HR of <80-110 beats/min is the management plan for a majority of patients who present to the ED in AF. According to the American Heart Association 2014 guidelines, the initial acute, emergent management of atrial fibrillation and flutter (AFF) are similar and there are a number of medications used for rate control including beta blockers and non-dihydropyridine calcium channel blockers.

Diltiazem, a non-dihydropyridine calcium channel blocker, is often the medication of choice in the management of AFF due to its ability to be given as an intravenous (IV) push, continuous infusion, and oral (PO) immediate release or extended release tablet. In the ED, a loading dose of IV diltiazem 0.25 mg/kg is usually administered to obtain a heart rate of < 110 beats/min or a decrease of at least 20% in the ventricular rate. If this does not work then a second bolus of 0.35mg/kg is administered. Once rate control of <110 beats/min or a 20% decrease in ventricular rate is obtained physicians typically chose between oral immediate release diltiazem tablet or IV continuous infusion diltiazem to maintain heart rate control. Both options allow for dose changes in the short term. The oral immediate release diltiazem tablet has a fast onset of action of 30-60 minutes and is dosed every 6 hours. Intravenous continuous infusion diltiazem has a variable onset of action with a titration frequency of every 15-30 minutes. The use of oral diltiazem allows for possible placement on a monitored general floor bed, whereas an intravenous drip requires placement to step down or intensive level of care. This impacts bed status and length of stay in the emergency department. Both oral and intravenous diltiazem are used clinically; however, no prospective studies exist comparing the two strategies. Retrospective data suggests that both forms are equal in their ability to control heart rate.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old
* Atrial fibrillation or flutter on electrocardiogram
* Heart rate >110 beats/min
* Systolic blood pressure >/= 90 mmHg

Exclusion Criteria:

* Limited English proficiency (LEP)
* Pregnant
* Prisoners
* Wolff Parkinson White syndrome
* Administration of electrical or chemical cardioversion before screening
* Administration of other antiarrhythmics for acute heart rate control (excluding adenosine)
* History of allergy or idiosyncratic reaction to diltiazem
* Unable to take oral medications
* Heart rate <60 beats/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy T Nguyen, PharmD, BCPS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Immediate Release Diltiazem | Continuous Infusion IV Diltiazem
Started | 9 | 10
Completed | 8 | 6
Not Completed | 1 | 4
Not completed — Treatment no longer indicated | 1 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Immediate Release Diltiazem | Continuous Infusion IV Diltiazem | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (11.6) | 58.3 (9.9) | 59.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Control
Description: Number of participant achieving heart rate control (defined as: HR <110 beats/min or conversion to sinus rhythm) at 2 hours after medication administration between oral immediate release and intravenous continuous infusion diltiazem
Time Frame: 2 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Immediate Release Diltiazem | Continuous Infusion IV Diltiazem
Number analyzed (Participants) | 8 | 6
Participants | 8 | 4

2. Secondary Outcome: Adverse Event Rate
Description: Number of participants with heart rate or blood pressure adverse events: Heart rate < 60 beats/min, or systolic blood pressure <90 mmHg requiring intervention (intravenous fluid bolus, vasopressors, medication discontinuation)
Time Frame: 4 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Immediate Release Diltiazem | Continuous Infusion IV Diltiazem
Number analyzed (Participants) | 8 | 6
Participants | 1 | 0

3. Other Pre Specified Outcome: Participant Specific Variables Associated With Heart Rate Control in Each Treatment Arm
Description: These variables include: Age, sex, race, weight, history of atrial fibrillation or flutter, history of hypertension, history of congestive heart failure, prior medication therapy, mean initial HR, duration of atrial fibrillation or flutter episode (<48 hrs or >48 hrs), mean initial diltiazem dose (mg/kg)
Time Frame: 4 hrs
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 hours
Description: self report by participant Only bradycardia (HR <60 beats/min) or hypotension (SBP <90 mmHg requiring intervention including IVF bolus administration, vasopressors, or medication discontinuation) related adverse events were recorded.
  Mortality was not recorded Non-serious adverse events were not recorded
Arm/Group | Oral Immediate Release Diltiazem | Continuous Infusion IV Diltiazem
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Immediate Release Diltiazem (N=8) | Continuous Infusion IV Diltiazem (N=6)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Braydcardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT03472495/Prot_SAP_000.pdf